CLINICAL TRIAL: NCT00993993
Title: Relational Development in Children With Cleft Lips and Palates: Influence of the Waiting Period Prior to the First Surgical Intervention and the Parents' Psychological Perception of the Abnormality
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 4506
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2015-09

CONDITIONS: Cleft Palate
Keywords: cleft palate
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- group "early intervention"
- group "late intervention"

SUMMARY:
The treatment of patients suffering from cleft lip(s) with or without a cleft palate (CL/P) is multidisciplinary. The careful consideration of concerned families during the repetitive appointments required by these treatments show the importance of the psychological context and of the harmonious structuring of the parents-child relationships on the child's development. Yet the birth of a child affected by CL/P is a particularly stressing and traumatising event for the parents. The investigators' prospective, multidisciplinary and multi-centred research project aims to assess the psychological perceptions of parents of children affected by CL/P over the year following the birth and analyse the child's degree of psychological suffering as well as the parents-child relationships. The time of the first surgical intervention varies amongst the treatment centres. The investigators listed four centres that intervene at different times according to the more or less long waiting times between the child's birth and this first surgical intervention. The results obtained for each group will be compared to one another and according to two sub-groups: parents who found out about the CL/P through embryo diagnosis and those who found out at their child's birth. The mental and psychological dimension due to the malformation and its correction will be analysed in the parents group (importance of the prenatal diagnosis, relational development with the child, self-esteem, quality of life) but also in the child (likely distress and withdrawal symptoms).

ELIGIBILITY:
Inclusion Criteria:

* Children with Cleft Lip with or without Cleft Palate and their Parents

Exclusion Criteria:

* Children with Cleft Palate without Cleft Lip
* Children born the 35th week of d'amenorrhea
* Children with a birth weight inferior to 1800 g
* Children put under care by court order
* Parents under administrative supervision
* Parents who are not familiar with the french language and/or illiterate

Ages: 4 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Primary care centers (France) Two referent centers Two competent centers
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-04-27 (Actual); Primary Completion 2010-04-27 (Actual); Study Completion 2013-01-07 (Actual)

PRIMARY OUTCOMES:
Assess the emotional state of withdrawal of any child carrying a CL/P based on the psychological state of their parents and time before the first surgery. We use ADBB scale for the child. | 2 years
Learning about the psychological effects of this abnormality on parents from the time of diagnosis and of the therapeutic management. We use PSI scale for the parents. | 2 years

SECONDARY OUTCOMES:
Indices of psychological distress by Quebec Health Survey (IDPESQ) and the Edinburgh Postnatal Depression Scale (EPDS).The Family Impact Scale. The Dyadic Adjustment Scale Spanier of determining the marital context and questionnaires ad-hoc. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: GROLLEMUND Bruno, MD, Principal Investigator — not affiliated
Locations (6):
- France (6):
  - CHRU, Centre de référence des malformations Cranio Maxillo Faciales Rares, Hôpital Salengro, Lille
  - CHU, Service de Chirurgie Maxillo-Faciale et Plastique de la Face Hôpital Central, Nancy
  - APHP Armand Trousseau, Centre de Référence des Malformations Rares de la Face et de la Cavité Buccale, Paris
  - CHRU, Service de Chirurgie Maxillo-Faciale Chirurgie B1, Strasbourg
  - CSERD, Pôle d'odontologie, Strasbourg
  - CHRU, Service de Chirurgie Infantile, Strasbourg

REFERENCES:
- [Derived] Perez Martinez C, Grollemund B, Gavelle P, Viaux-Savelon S, Guedeney A. The Prevalence of Social Withdrawal in Infants With Cleft Lip and Palate: The Feasibility of the Full and the Modified Versions of the Alarm Distress Baby Scale. Front Pediatr. 2022 Jul 7;10:804802. doi: 10.3389/fped.2022.804802. eCollection 2022. PMID 35874558
- [Derived] Grollemund B, Dissaux C, Gavelle P, Martinez CP, Mullaert J, Alfaiate T, Guedeney A; CLIP team (Cleft Lip & palate Infant Parent). The impact of having a baby with cleft lip and palate on parents and on parent-baby relationship: the first French prospective multicentre study. BMC Pediatr. 2020 May 18;20(1):230. doi: 10.1186/s12887-020-02118-5. PMID 32423402
- [Derived] Grollemund B, Guedeney A, Vazquez MP, Picard A, Soupre V, Pellerin P, Simon E, Velten M, Dissaux C, Kauffmann I, Bruant-Rodier C, Danion-Grilliat A. Relational development in children with cleft lip and palate: influence of the waiting period prior to the first surgical intervention and parental psychological perceptions of the abnormality. BMC Pediatr. 2012 Jun 8;12:65. doi: 10.1186/1471-2431-12-65. PMID 22682069